CLINICAL TRIAL: NCT06889116
Title: Correlation of Point of Care Venous Excess Ultrasonography (VExUS) Score and Acute Kidney Injury (AKI) in Critically Ill Adult Patients- a Prospective Observational Study.
Brief Title: VExUS Score and AKI in Critically Ill Adult patients-a Prospective Observational Study.
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Bipin Karki, Principle investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 438(6-11)E2- 079/080
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Acute Kidney Injury; VExUS
Keywords: VExUS; Acute Kidney Injury; Cumulative fluid balance; Point of Care Ultrasound
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with AKI: Patients who are admitted with the diagnosis of AKI or develop AKI during their ICU stay

SUMMARY:
Introduction Renal perfusion is dependent on the renal perfusion pressure across the renal capillaries. Venous congestion due to excess fluid therapy can drastically reduce the renal perfusion pressure in spite of a normal mean arterial pressure. Increasing cumulative fluid balance during the ICU stay has been found to be associated with negative outcomes including acute kidney injury (AKI) and hospital mortality. Venous excess ultrasound (VExUS) to assess the Doppler studies of renal, hepatic and portal veins along with the inferior venacava has been shown to reliably predict the incidence of AKI in certain ICU patient population more specifically in cardiorenal syndrome. The aim of this study was to correlate the incidence of AKI and VExUS scores in a mixed ICU population and hence determine the contribution of venous congestion on the causation of AKI in a general ICU.

Methods:

The patients included who have AKI at admission or developed AKI during their ICU stay were included. The definition of AKI used for this study was as defined by Kidney Disease: Improving Global Outcomes (KDIGO). Point of care VExUS scans were done on each patient at inclusion (day 0), then each day for a total of 4 days (day 1, 2 and 3), till initiation of renal replacement therapy, death or discharge form the ICU. Correlation between VExUS grades and creatinine clearances was explored as the primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Admitted to the adult ICUs of TUTH (ICU A and ICU B)
* Admitting diagnosis of AKI or who developed AKI during their ICU stay

Exclusion Criteria:

* Pregnancy
* Diagnosed case of chronic kidney disease
* Diagnosed case of cirrhosis/ portal hypertension
* Arrhythmias which would interfere with the acquisition and interpretation of the Doppler waveforms
* Inferior venacava thrombus
* Poor window for assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had AKI at the time of admission or who developed AKI during their ICU stay were screened for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
To determine correlation between the VExUS score with creatinine clearance. | At the end of Day 3 or initiation of renal replacement therapy or resolution of AKI, death or discharge from the ICU. whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan University Teaching Hospital, Mahārājgañj, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided